CLINICAL TRIAL: NCT02789189
Title: Nedaplatin Combined With Gemcitabine in the Treatment of Recurrent and/or Metastatic Nasopharyngeal Carcinoma : a Single Arm and Phase Ⅱ Clinical Trail
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Qingqing Cai, Professor, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: B2015-073-01
Record Dates: First submitted 2016-05-29; First posted 2016-06-02 (Estimated); Last update posted 2019-09-06 (Actual); Status verified 2016-05

CONDITIONS: Recurrent and Metastatic Nasopharyngeal Carcinoma
MeSH Terms: conditions — Recurrence; Nasopharyngeal Carcinoma | interventions — nedaplatin; Gemcitabine

ARMS (1):
- nedaplatin combined with gemcitabine (Experimental)
  Interventions: Drug: nedaplatin and gemcitabine

INTERVENTIONS:
Drug: nedaplatin and gemcitabine

SUMMARY:
The purpose of this single arm,phase Ⅱ clinical trail is to determine the safety and efficacy of nedaplatin combined with gemcitabine in the treatment of recurrent and metastatic nasopharyngeal carcinoma

ELIGIBILITY:
Inclusion Criteria:

* biopsy proved nasopharyngeal carcinoma; stage IVc according to Union for International Cancer Control (UICC) edition VII,or recurrent disease after chemotherapy and/or radiotherapy; 18 years or older; without other malignancy; proper functioning of the major organs.

Exclusion Criteria:

* allergic to nedaplatin and/or gemcitabine; female within gestation period or lactation; patients received drug of other clinical trail within 3 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2016-06; Primary Completion 2019-09-04 (Actual)

PRIMARY OUTCOMES:
overall survival | 5 years